CLINICAL TRIAL: NCT02472028
Title: LEukoaraiosis and blOod Pressure Reduction in OLD People
Brief Title: Blood Pressure Reduction to Limit the Evolution of Vascular Brain Lesions in Elderly Individuals
Acronym: LEOPOLD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P100153; 2014 A00265-42 (Other: IDRCB)
Record Dates: First submitted 2015-04-27; First posted 2015-06-15 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Cerebrovascular Disorders
Keywords: Cerebrovascular Disorders; Stroke; Antihypertensive Agents; Arterial Pressure; Memory Disorders
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- blood pressure lowering algorithm (Experimental): enhanced strategy aiming to reduce systolic blood pressure to <135 mmHg
  Interventions: Other: blood pressure lowering algorithm
- usual strategy (Active Comparator): usual strategy based on the usual care of routine care
  Interventions: Other: usual strategy

INTERVENTIONS:
Other: blood pressure lowering algorithm — The treatments used in the "enhanced strategy" arm are those proposed by national (HAS2013, SFHTA2013) and international (ESH 2013) recommendations, according to their Marketing Authorization and Summary of Product Characteristics : Diuretics, beta-blockers, Angiotensin Converting Enzyme inhibitors, Angiotensin Receptor Blockers, Calcium Channel Blockers Throughout the study, choice of drugs in each therapeutic class is left on the investigator's initiative. All drugs of these classes may be used , no specific drug is tested in this study.
  Other Names: enhanced strategy
  Arms: blood pressure lowering algorithm
Other: usual strategy — The implementation of antihypertensive therapy the current recommendations to reach the blood pressure target in usual care. Throughout the study, choice of drugs in each therapeutic class is left on the investigator's initiative. Combinations of different pharmacological classes can be tested in order to find the most effective and best tolerated combinations.
  Arms: usual strategy

SUMMARY:
The purpose of the study is to test the hypothesis of slowing the progression of White Matter Lesions (WML) by lowering blood pressure (BP) in patients with cognitive complaints and a moderate to high grade of WML on brain MRI.

DETAILED DESCRIPTION:
SCIENTIFIC BACKGROUND: White Matter Lesions (WML) are cerebrovascular abnormalities discovered on MRI that are associated with an increased risk of dementia. High blood pressure (BP) is a major risk factor for WML. WML are therefore key lesions in the causal chain linking vascular factors and dementia, particularly Alzheimer's disease.

However, it has not been shown that lowering BP could limit the progression of the WML in people with cognitive impairment.

OBJECTIVES: To test the hypothesis of slowing progression of WML by lowering BP in patients with memory complaints with a moderate to high grade of WML on brain MRI.

STUDY DESIGN: PROBE (Prospective randomized open blinded end-point) trial. Blind reading of both MRI for every patient in each group. After stratified randomization on age, sex and center, patients will be assigned to two strategies:

* Reinforced Group (RG): enhanced strategy aiming at a systolic BP <135 mmHg;
* Usual Group (UG): usual strategy based on the usual routine care.

SAMPLE SIZE: patients will be enrolled (410 in each arm) in 12 Memory Resources and Research Center (CMRR) with access to 1.5 T or more MRI.

CONDUCT OF THE STUDY:

Duration of the inclusion period: 96 months and 2 weeks. Patient participation duration: 36 months + 6 months max Total study duration: 11 years. Clinical and para-clinical evaluation: MRI as part of research at the beginning of the study and before the end of the study at 36 months + 6 months max (primary endpoint); Clinical evaluation of neuropsychological tests at the beginning of the study and yearly ; walking speed measurement single leg stance balance test ; repeated BP measurements; monitoring of neurological signs and symptoms; blood test at the beginning of the study (electrolytes, lipid profiles, fasting blood glucose, if not existing); MRI if not existing for validation of the inclusion criterion and performed in the ordinary course.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 88 years old patients;
* Patient with cognitive complaint with MMSE ≥ 20performed within 6 months prior to enrollment (with or without dementia)
* Patient with a socio-educational level ≥ 3
* Presence of hyperintensities of moderate to high grade on the last MRI or old scan (grades C and D on the modified Scheltens scale, grades 2/3 Fazekas).
* Hypertension defined by a Systolic Blood Pressure (SBP) and / or a Diastolic Blood Pressure (DBP) ≥ 140/90 mmHg, treated or not
* Affiliation to a social security system
* Informed consent given, signed consent

Exclusion Criteria:

* Presence of severe orthostatic hypotension defined as a decrease of 30 mmHg in SBP standing within 3 minutes
* Contraindication to MRI (presence of ferromagnetic foreign body (especially some intracranial clips, some heart valves, intraocular foreign bodies, metal prosthesis), subject carrying pacemaker, claustrophobic participants)
* Severe diseases associated with a life expectancy of less than 3 months;
* Major physical impairments that can interfere with the feasibility of the tests (sight, hearing ...)
* Presence of another dementia different than Alzheimer's disease vascular dementia or mixed dementia,
* Persons under guardianship;
* Secondary hypertension: renovascular hypertension, primary aldosteronism, pheochromocytoma ...;
* Patient already receiving 4 or more antihypertensive drugs at maximum dosage
* Patient participating in another clinical research study on drug requiring exclusion period
* severe renal impairment

Ages: 60 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2028-09-11 (Estimated); Study Completion 2028-09-11 (Estimated)

PRIMARY OUTCOMES:
The main criterion is based on the quantitative assessment of White Matter Lesions (WML) volumes at the beginning and at the end of the study for each patient and each arm of the trial. The WML volume from the final MRI is compared to that of the initial | 36 months + 6 months max

SECONDARY OUTCOMES:
Imaging criteria : changes in the number of large or confluent WML | 36 months+ 6 months max
Imaging criteria : changes in the volume of WML depending on their location (periventricular and deep white matter) | 36 months+ 6 months max
Imaging criteria : changes in the number of silent infarctus | 36 months+ 6 months max
Imaging criteria : changes in the number of microbleeds | 36 months+ 6 months max
Imaging criteria : evolution of brain volumes (gray matter, white matter, CSF, and regional volumes including hippocampus) | 36 months+ 6 months max
Clinical criteria: clinical criteria (changes in neuropsychological tests | 36 months
Clinical criteria: changes inwalking speed | 36 months
Clinical criteria: number of incident cases of dementia | 36 months
Number of incident cases of vascular events validated by an expert committee | 36 months
Clinical criteria: total mortality by cause | 36 months+ 6 months max

CONTACTS AND LOCATIONS:
Overall Officials: Christophe TZOURIO, MD, PhD, Study Director — Inserm U897 - Bordeaux University; Olivier HANON, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Memory for Research and Resources Center / Neuroscience pole, Bordeaux, Pellegrin Hospital Group
  - Memory Resources Centre and South of Ile de France Search - Broca Hospital, Paris